CLINICAL TRIAL: NCT06588374
Title: The Effect of Lateral Internal Sphincterotomy During Hemorrhoidectomy ,a Randomized Clinical Trial.
Brief Title: Hemorrhoidectomy Only Versus Hemorrhoidectomy With Lateral Internal Sphincterotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mohamed Ahmed, Resident Doctor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hemorrhoidectomy
Record Dates: First submitted 2024-02-26; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Lateral Internal Sphincterotomy

STUDY DESIGN:
Intervention Model Description: hemorrhoidectomy alone versus hemorrhoidectomy with lateral internal sphincterotomy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemorrhoidectomy Only (Experimental): Hemorrhoids by Hemorrhoidectomy alone
  Interventions: Procedure: lateral internal sphincterotomy
- Hemorrhoidectomy With Lateral Internal Sphincterotomy (Experimental): hemorroids by lateral internal sphincterotomy and hemorrhoidectomy
  Interventions: Procedure: lateral internal sphincterotomy

INTERVENTIONS:
Procedure: lateral internal sphincterotomy — Hemorrhoidectomy versus Hemorrhoidectomy with lateral internal sphincterotomy

SUMMARY:
The aim of this study was to access the comparison of pain and complications after hemorrhoidectomy with or without lateral sphincterotomy.

DETAILED DESCRIPTION:
Hemorrhoids arise from congestion of anal cushions and characteristically lie in the 3, 7 and 11 O clock positions (with the patient in lithotomy position) . The most common complication of open hemorrhoidectomy is postoperative pain caused by spasm of the internal sphincter . Lateral internal sphincterotomy is one good technique. It reduces pain by reducing spasm of internal anal sphincter which is the main cause of pain . The addition of lateral internal sphincterotomy to haemorrhoidectomy resulted in generally lower postoperative anal pressures . The long-term outcomes, which included anal stenosis and anal fissure, were significantly lower after lateral internal sphincterotomy . patients with recurrence of hemorrhoids, severe pain, prolonged constipation, or anyone with high sphincter tonicity in the digital rectal examination would be a candidate for manometric evaluation of anal canal pressure. These patients with high analcanal pressure confirmed with manometry might receive internal sphincterotomy plus hemorrhoid-ectomy .

ELIGIBILITY:
Inclusion Criteria:

1. Surgically fit according to ASA.
2. Cases with hemorrhoids Grade ll& III & IV.
3. Age between (18-60).

Exclusion Criteria:

1. Age less than 18 years old.
2. Complete rectal prolapse.
3. Grade I hemorrhoids.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Effect of Hemorrhoidectomy versus Hemorrhoidectomy with lateral internal sphincterotomy on post operative complications | Baseline
  To assess postoperative pain intensity by Numberical rating scale 0 To 10

CONTACTS AND LOCATIONS:
Overall Officials: ashraf A Helmy, professor, Principal Investigator — Assiut University

REFERENCES:
- See also: The Role of Lateral Internal Sphincterotomy in Haemorrhoidectomy: A Study in a Tertiary Care Center — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8277982/
- See also: Comparison of hemorrhoidectomy combined with LIS and open hemorrhoidectomy — https://theprofesional.com/index.php/tpmj/article/view/4580
- See also: Randomized controlled trial of lateral internal sphincterotomy with haemorrhoidectomy — https://pubmed.ncbi.nlm.nih.gov/8665199/
- See also: The Role of Lateral Internal Sphincterotomy in Haemorrhoidectomy: A Study in a Tertiary Care Center — https://pubmed.ncbi.nlm.nih.gov/34306842/